CLINICAL TRIAL: NCT04911218
Title: Randomized Comparison of GlideSheath Slender® Versus Conventional 5Fr Arterial Sheath in Coronary Angiography Through the Distal Radial Artery (Anatomical Snuffbox)
Brief Title: GlideSheath Slender® Versus Conventional 5Fr Arterial Sheath in Coronary Angiography Through the Distal Radial Artery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Grigorios Tsigkas, Assistant Professor of Cardiology, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1762/22.01.21
Record Dates: First submitted 2021-05-20; First posted 2021-06-02 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Arterial Access; Coronary Angiography; Radial Artery Occlusion
Keywords: arterial access; coronary angiography; radial access; distal radial access; radial artery occlusion
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GlideSheath Slender 5Fr arterial sheath (Experimental): Placement of GlideSheath Slender 5Fr arterial sheath for diagnostic angiography through the distal radial artery (anatomical snuffbox).
  Interventions: Device: GlideSheath Slender 5Fr arterial sheath
- Conventional 5Fr arterial sheath (Active Comparator): Placement of Conventional 5Fr arterial sheath arterial sheath for diagnostic angiography through the distal radial artery (anatomical snuffbox).
  Interventions: Device: Conventional 5Fr arterial sheath

INTERVENTIONS:
Device: GlideSheath Slender 5Fr arterial sheath — Placement of GlideSheath Slender 5Fr arterial sheath for coronary angiography through the distal radial artery (anatomical snuffbox).
  Arms: GlideSheath Slender 5Fr arterial sheath
Device: Conventional 5Fr arterial sheath — Placement of conventional 5Fr arterial sheath for coronary angiography through the distal radial artery (anatomical snuffbox).
  Arms: Conventional 5Fr arterial sheath

SUMMARY:
Transradial approach has become the default arterial access for coronary angiography (CAG) and percutaneous coronary intervention (PCI), mainly due to lower incidence of bleeding compared to transfemoral access.1 However, TRA is not deprived of local access site complications such as radial artery occlusion (RAO), occurring in approximately 5.2% of patients, compartment syndrome, pseudoaneurysm, hematoma, and arteriovenous fistula. Recently, a novel approach has been proposed, the access through the distal radial artery (distal transradial access, dTRA), located in the anatomical snuffbox. Initial studies regarding the dRA have shown feasibility and benefits, including shorter hemostasis time, fewer local access site complications and potentially lower incidence of RAO.

GlideSheath Slender is a novel sheath which has a hydrophilic coating and is made of a thinner material than traditional sheaths. As a result, the external diameter of the 5 Fr GlideSheath Slender sheath is 1 Fr lower compared with conventional arterial sheaths.

The purpose of the present study was to investigate whether the use of the Slender sheath affects the time of hemostasis, sheath insertion time, crossover rate to conventional radial access, pain associated with the procedure and incidence of local access site complications (RAO, distal radial artery occlusion, fistula, hematoma) in patients undergoing diagnostic angiography through the distal radial artery.

DETAILED DESCRIPTION:
Patients fulfilling the enrollment criteria will be randomized 1:1 to GlideSheath Slender versus conventional 5Fr arterial sheath for access through the distal radial artery (dTRA). In case an interventional procedure is required then the initial sheath will be exchanged to a larger sheath according to the circumstances of the case and the patient will not be included in the analysis.

For randomized patients sheath insertion time, necessity for crossover to conventional radial access, pain associated with the procedure (visual pain scale) and occurrence of hematoma will be recorded. Follow-up ultrasound 7-10 days after the procedure for detection of RAO, distal radial artery occlusion and fistula formation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Indication for coronary angiography
* Age>18 years
* Informed consent

Exclusion Criteria:

* Non-palpable right radial artery
* Prior CABG
* STEMI
* Prior right transaradial intervention within the previous 2 months
* Hemodynamic instability
* Anatomical restrictions (fistula orthopaedic problems, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-11-25 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
Rate of successful hemostasis at 30 minutes after sheath removal | At 30 minutes after sheath removal

SECONDARY OUTCOMES:
Crossover rate to conventional radial access | During the procedure
Pain associated with the procedure (visual analog scale, VAS) | During the procedure
  0-10, 0: no pain, 10: worst pain possible
Rate of hematoma modified EASY class≥II | Up to 24 hours after hemostatic device removal
Rate of forearm radial artery occlusion | 7-10 days after the coronary angiography
Rate of distal radial artery occlusion | 7-10 days after the coronary angiography
Rate of fistula formation | 7-10 days after the coronary angiography
Rate of pseudoaneurysm formation | 7-10 days after the coronary angiography

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece

IPD SHARING:
Plan to Share IPD: No